CLINICAL TRIAL: NCT02001623
Title: First-in-human, Dose-escalating Safety Study of Tissue Factor Specific Antibody Drug Conjugate Tisotumab Vedotin (HuMax® TF ADC) in Patients With Locally Advanced and/or Metastatic Solid Tumors Known to Express Tissue Factor
Brief Title: Tisotumab Vedotin (HuMax®-TF-ADC) Safety Study in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Collaborators: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GEN701; innovaTV 201 (Other: Genmab)
Record Dates: First submitted 2013-11-14; First posted 2013-12-05 (Estimated); Results first posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-11

CONDITIONS: Ovary Cancer; Cervix Cancer; Endometrium Cancer; Bladder Cancer; Prostate Cancer (CRPC); Esophagus Cancer; Lung Cancer(NSCLC); Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Keywords: ovary cancer; cervix cancer; endometrium cancer; bladder cancer; prostate cancer (CRPC); esophagus cancer; lung cancer(NSCLC); Squamous cell carcinoma of the head and neck (SCCHN)
MeSH Terms: conditions — Ovarian Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Urinary Bladder Neoplasms; Prostatic Neoplasms; Esophageal Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — tisotumab vedotin

STUDY DESIGN:
Intervention Model Description: Escalation phase for dose finding followed by expansion phase
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- Tisotumab Vedotin (HuMax-TF-ADC) (Experimental): All arms of the trial (borh in escalation and expansion phase) will be administered tisotumab vedotin (HuMax-TF-ADC)
  Interventions: Drug: Tisotumab Vedotin (HuMax-TF-ADC)

INTERVENTIONS:
Drug: Tisotumab Vedotin (HuMax-TF-ADC)
  Other Names: TIVDAK

SUMMARY:
The purpose of the trial is to establish the tolerability of HuMax-TF-ADC in a mixed population of patients with specified solid tumors.

DETAILED DESCRIPTION:
The study is conducted in two parts. The dose escalation portion of the trial subjects are enrolled into cohorts at increasing dose levels of HuMax-TF-ADC in 21 day treatment cycles.

In the Cohort Expansion part of the trial, will further explore the recommended phase 2 dose of HuMax-TF-ADC as determined in Part 1

ELIGIBILITY:
Inclusion Criteria:

- Patients with relapsed, advanced and/or metastatic cancer who have failed available standard treatments or who are not candidates for standard therapy.

Patients must have measurable disease

* Age ≥ 18 years.
* Acceptable renal function
* Acceptable liver function
* Acceptable hematological status (without hematologic support
* Acceptable coagulation status
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy of at least three months.
* A negative serum pregnancy test (if female and aged between 18-55 years old).
* Women who are pregnant or breast feeding are not to be included.
* Patients, both females and males, of reproductive potential must agree to use adequate contraception during and for six months after the last infusion of HuMax-TF-ADC.
* Following receipt of verbal and written information about the study, patients must provide signed informed consent before any study-related activity is carried out.

Exclusion Criteria:

* Known past or current coagulation defects.
* Ongoing major bleeding,
* Have clinically significant cardiac disease
* A baseline QT interval as corrected by Fridericia's formula (QTcF) > 450 msec, a complete left bundle branch block (defined as a QRS interval ≥ 120 msec in left bundle branch block form) or an incomplete left bundle branch block.
* Have received granulocyte colony stimulating factor (G-CSF) or granulocyte/macrophage colony stimulating factor support within one week or pegylated G-CSF within two weeks before the Screening Visit.
* Have received a cumulative dose of corticosteroid ≥ 100 mg (prednisone or equivalent doses of corticosteroids) within two weeks before the first infusion.
* Major surgery within six weeks or open biopsy within 14 days before drug infusion.
* Plan for any major surgery during treatment period.
* Any history of intracerebral arteriovenous malformation, cerebral aneurysm, brain metastases or stroke.
* Any anticancer therapy including; small molecules, immunotherapy, chemotherapy monoclonal antibodies or any other experimental drug within four weeks or five half lives, whichever is longest, before first infusion.
* Prior treatment with bevacizumab within twelve weeks before the first infusion.
* Radiotherapy within 28 days prior to first dose.
* Patients who have not recovered from symptomatic side effects of radiotherapy at the time of initiation of screening procedure.
* Known past or current malignancy other than inclusion diagnosis, except for:
* Cervical carcinoma of Stage 1B or less.
* Non-invasive basal cell or squamous cell skin carcinoma.
* Non-invasive, superficial bladder cancer.
* Prostate cancer with a current PSA level < 0.1 ng/mL.
* Any curable cancer with a complete response (CR) of > 5 years duration.
* Known human immunodeficiency virus seropositivity.
* Positive serology (unless due to vaccination or passive immunization due to Ig therapy) for hepatitis B
* Positive serology for hepatitis C based on test at screening.
* Inflammatory bowel disease including Crohn's disease and colitis ulcerosa.
* Inflammatory lung disease including moderate and severe asthma and chronic obstructive pulmonary disease (COPD) requiring chronic medical therapy.
* Ongoing acute or chronic inflammatory skin disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2013-11-30 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2019-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johann de Bono, Professor, Principal Investigator — The Institute of Cancer Research & The Royal Marsden NHS Foundation Trust
Locations (29):
- United States (8):
  - University of California Irvine Medical Center (UCIMC), Orange, California
  - Yale Cancer Center, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - University Gynecologic Oncology, Atlanta, Georgia
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
- Belgium (8):
  - Universitair Ziekenhuis Antwerpen, Edegem, Antwerpen
  - Universitair Ziekenhuis Leuven, Leuven, Flemish Brabant
  - Grand Hôpital de Charleroi, Charleroi, Hainaut
  - Centre Hospitalier Universitaire Ambroise Paré, Mons, Hainaut
  - CHU UCL Namur - site Godinne, Yvoir, Namur
  - Saint-Luc University Hospital, Brussels
  - CHU de Liège, Liège
  - CHU UCL Namur - Sainte Elisabeth, Namur
- Denmark (2):
  - Rigshospitalet, Copenhagen University Hospital, Copenhagen
  - Herlev and Gentofte Hospital, Herlev
- Sweden (2):
  - Karolinska Universitetssjukhuset, Stockholm, Solna
  - Lungemedicinska Kliniken, Linköping
- United Kingdom (9):
  - The Leeds Teaching Hospitals NHS Trust, Leeds, England
  - University College London Hospitals, London, England
  - Sarah Cannon Research Institute - London, London, England
  - Newcastle Hospitals NHS Foundation Trust, Newcastle upon Tyne, Newcastle
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - Velindre NHS Trust, Cardiff, Wales
  - Beatson Cancer Centre, Glasgow
  - Guys hospital, London
  - The Christie NHS Foundation Trust, Manchester

REFERENCES:
- [Result] de Bono JS, Concin N, Hong DS, Thistlethwaite FC, Machiels JP, Arkenau HT, Plummer R, Jones RH, Nielsen D, Windfeld K, Ghatta S, Slomovitz BM, Spicer JF, Yachnin J, Ang JE, Mau-Sorensen PM, Forster MD, Collins D, Dean E, Rangwala RA, Lassen U. Tisotumab vedotin in patients with advanced or metastatic solid tumours (InnovaTV 201): a first-in-human, multicentre, phase 1-2 trial. Lancet Oncol. 2019 Mar;20(3):383-393. doi: 10.1016/S1470-2045(18)30859-3. Epub 2019 Feb 8. PMID 30745090
- [Derived] Feng S, Gunawan R, Passey C, Voellinger J, Polhamus D, Gerritsen A, O'Day C, Carret AS, Soumaoro I, Gupta M, Hanley WD. Exposure-safety Markov modeling of ocular adverse events in patient populations treated with tisotumab vedotin. J Pharmacokinet Pharmacodyn. 2025 Oct 3;52(5):55. doi: 10.1007/s10928-025-10003-w. PMID 41044356
- [Derived] Passey C, Voellinger J, Gibiansky L, Gunawan R, Nicacio L, Soumaoro I, Hanley WD, Winter H, Gupta M. Exposure-safety and exposure-efficacy analyses for tisotumab vedotin for patients with locally advanced or metastatic solid tumors. CPT Pharmacometrics Syst Pharmacol. 2023 Sep;12(9):1262-1273. doi: 10.1002/psp4.13007. Epub 2023 Jul 26. PMID 37496366
- [Derived] Hong DS, Concin N, Vergote I, de Bono JS, Slomovitz BM, Drew Y, Arkenau HT, Machiels JP, Spicer JF, Jones R, Forster MD, Cornez N, Gennigens C, Johnson ML, Thistlethwaite FC, Rangwala RA, Ghatta S, Windfeld K, Harris JR, Lassen UN, Coleman RL. Tisotumab Vedotin in Previously Treated Recurrent or Metastatic Cervical Cancer. Clin Cancer Res. 2020 Mar 15;26(6):1220-1228. doi: 10.1158/1078-0432.CCR-19-2962. Epub 2019 Dec 3. PMID 31796521

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In the dose escalation part of the study, 40 participants were screened and 27 were enrolled and received treatment. In the dose expansion part of the study, 294 participants were screened and 168 were enrolled and received treatment.
Groups:
- Dose Escalation Part: 0.3 mg/kg: Participants received tisotumab vedotin on Day 1 of each cycle (each treatment cycle was 21 days) as an intravenous (IV) infusion at a dose of 0.3 mg/kg of body weight.
- Dose Escalation Part: 0.6 mg/kg: Participants received tisotumab vedotin on Day 1 of each cycle (each treatment cycle was 21 days) as an IV infusion at a dose of 0.6 mg/kg of body weight.
- Dose Escalation Part: 0.9 mg/kg: Participants received tisotumab vedotin on Day 1 of each cycle (each treatment cycle was 21 days) as an IV infusion at a dose of 0.9 mg/kg of body weight.
- Dose Escalation Part: 1.2 mg/kg: Participants received tisotumab vedotin on Day 1 of each cycle (each treatment cycle was 21 days) as an IV infusion at a dose of 1.2 mg/kg of body weight.
- Dose Escalation Part: 1.5 mg/kg: Participants received tisotumab vedotin on Day 1 of each cycle (each treatment cycle was 21 days) as an IV infusion at a dose of 1.5 mg/kg of body weight.
- Dose Escalation Part: 1.8 mg/kg: Participants received tisotumab vedotin on Day 1 of each cycle (each treatment cycle was 21 days) as an IV infusion at a dose of 1.8 mg/kg of body weight.
- Dose Escalation Part: 2.0 mg/kg: Participants received tisotumab vedotin on Day 1 of each cycle (each treatment cycle was 21 days) as an IV infusion at a dose of 2.0 mg/kg of body weight.
- Dose Escalation Part: 2.2 mg/kg: Participants received tisotumab vedotin on Day 1 of each cycle (each treatment cycle was 21 days) as an IV infusion at a dose of 2.2 mg/kg of body weight.
- Dose Expansion Part: Bladder Cancer: Participants with bladder cancer received tisotumab vedotin on Day 1 of each cycle (each treatment cycle was 21 days) as an IV infusion at a dose of 2.0 mg/kg of body weight.
- Dose Expansion Part: Cervical Cancer: Participants with cervical cancer received tisotumab vedotin on Day 1 of each cycle (each treatment cycle was 21 days) as an IV infusion at a dose of 2.0 mg/kg of body weight.
- Dose Expansion Part: Endometrial Cancer: Participants with endometrial cancer received tisotumab vedotin on Day 1 of each cycle (each treatment cycle was 21 days) as an IV infusion at a dose of 2.0 mg/kg of body weight.
- Dose Expansion Part: Esophageal Cancer: Participants with esophageal cancer received tisotumab vedotin on Day 1 of each cycle (each treatment cycle was 21 days) as an IV infusion at a dose of 2.0 mg/kg of body weight.
- Dose Expansion Part: Non-Small Cell Lung Cancer (NSCLC): Participants with NSCLC received tisotumab vedotin on Day 1 of each cycle (each treatment cycle was 21 days) as an IV infusion at a dose of 2.0 mg/kg of body weight.
- Dose Expansion Part: Ovarian Cancer: Participants with ovarian cancer received tisotumab vedotin on Day 1 of each cycle (each treatment cycle was 21 days) as an IV infusion at a dose of 2.0 mg/kg of body weight.
- Dose Expansion Part: Prostate Cancer: Participants with prostate cancer received tisotumab vedotin on Day 1 of each cycle (each treatment cycle was 21 days) as an IV infusion at a dose of 2.0 mg/kg of body weight.
Period: Overall Study
Arm/Group | Dose Escalation Part: 0.3 mg/kg | Dose Escalation Part: 0.6 mg/kg | Dose Escalation Part: 0.9 mg/kg | Dose Escalation Part: 1.2 mg/kg | Dose Escalation Part: 1.5 mg/kg | Dose Escalation Part: 1.8 mg/kg | Dose Escalation Part: 2.0 mg/kg | Dose Escalation Part: 2.2 mg/kg | Dose Expansion Part: Bladder Cancer | Dose Expansion Part: Cervical Cancer | Dose Expansion Part: Endometrial Cancer | Dose Expansion Part: Esophageal Cancer | Dose Expansion Part: Non-Small Cell Lung Cancer (NSCLC) | Dose Expansion Part: Ovarian Cancer | Dose Expansion Part: Prostate Cancer
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 15 | 55 | 14 | 15 | 15 | 36 | 18
Completed 4 Cycles of Treatment | 0 | 1 | 1 | 2 | 0 | 2 | 2 | 1 | 5 | 31 | 6 | 4 | 6 | 22 | 7
Completed 12 Cycles of Treatment | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 0
Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0
Not Completed | 3 | 3 | 3 | 2 | 3 | 3 | 3 | 6 | 15 | 53 | 14 | 15 | 14 | 35 | 18
Not completed — Disease Progression | 2 | 2 | 3 | 2 | 3 | 2 | 3 | 3 | 7 | 40 | 5 | 9 | 9 | 20 | 9
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 3 | 3 | 1 | 2 | 1
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 4 | 6 | 4 | 0 | 3 | 5 | 6
Not completed — Other - Miscellaneous | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 2 | 1 | 5 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Start of New Anti-cancer Treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Dose Delay Due to Toxicity | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set: all participants who had been exposed to tisotumab vedotin in either the dose escalation or expansion parts.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Part: 0.3 mg/kg | Dose Escalation Part: 0.6 mg/kg | Dose Escalation Part: 0.9 mg/kg | Dose Escalation Part: 1.2 mg/kg | Dose Escalation Part: 1.5 mg/kg | Dose Escalation Part: 1.8 mg/kg | Dose Escalation Part: 2.0 mg/kg | Dose Escalation Part: 2.2 mg/kg | Dose Expansion Part: Bladder Cancer | Dose Expansion Part: Cervical Cancer | Dose Expansion Part: Endometrial Cancer | Dose Expansion Part: Esophageal Cancer | Dose Expansion Part: Non-Small Cell Lung Cancer (NSCLC) | Dose Expansion Part: Ovarian Cancer | Dose Expansion Part: Prostate Cancer | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 15 | 55 | 14 | 15 | 15 | 36 | 18 | 195
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Preterm newborn infants (gestational age < 37 wks) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Children (2-11 years) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Adolescents (12-17 years) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Adults (18-64 years) | 3 | 1 | 3 | 3 | 2 | 2 | 2 | 4 | 12 | 51 | 8 | 8 | 9 | 26 | 4 | 138
  From 65-84 years | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 2 | 3 | 4 | 6 | 7 | 6 | 10 | 14 | 57
  85 years and over | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 2 | 2 | 3 | 3 | 5 | 2 | 55 | 14 | 3 | 12 | 36 | 0 | 140
  Male | 2 | 2 | 2 | 1 | 1 | 0 | 0 | 1 | 13 | 0 | 0 | 12 | 3 | 0 | 18 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
  Not Hispanic or Latino | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 15 | 53 | 13 | 15 | 15 | 35 | 18 | 191
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 15 | 49 | 14 | 13 | 13 | 34 | 17 | 182
  Black or Asian American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 1 | 0 | 0 | 5
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
  Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Dose Escalation Part: Evaluation of Treatment-Emergent Adverse Events
Description: Evaluation of treatment-emergent adverse events (TEAEs) includes number of participants with at least one:
  TEAE Serious TEAE Infusion-related TEAE Common Terminology Criteria for Adverse Events (CTCAE) grade >=3 Treatment-related TEAE
  A CTCAE TEAE was determined using the CTCAE grading systems based on National Cancer Institute (NCI)-CTCAE version 4.03 assessed by the investigator per the below definitions.
  Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living.
  Grade 4: Life-threatening consequences; urgent intervention indicated. Grade 5: Death related to AE.
Time Frame: Treatment emergent adverse events are reported from Day 1 to 30 days after dosing. The treatment duration ranged from 1 to 249 days in the dose escalation part.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Part: 0.3 mg/kg | Dose Escalation Part: 0.6 mg/kg | Dose Escalation Part: 0.9 mg/kg | Dose Escalation Part: 1.2 mg/kg | Dose Escalation Part: 1.5 mg/kg | Dose Escalation Part: 1.8 mg/kg | Dose Escalation Part: 2.0 mg/kg | Dose Escalation Part: 2.2 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6
Participants
  TEAEs | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6
  Serious TEAEs | 2 | 1 | 0 | 2 | 2 | 2 | 2 | 4
  Infusion-Related TEAEs | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CTCAE Grade >=3 TEAEs | 2 | 3 | 1 | 1 | 2 | 3 | 2 | 4
  TEAEs Related to Study Drug | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 6

2. Secondary Outcome: Dose Escalation and Expansion Part: Number of Participants With Markedly Abnormal Hematology Values
Description: Number of participants with markedly abnormal hematology values was defined as all participants who experienced at least 1 CTCAE grade >= 3 hematology value.
  A markedly abnormal hematology value was determined using the CTCAE grading systems based on National Cancer Institute (NCI)-CTCAE version 4.03 assessed by the investigator per the below definitions.
  Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living.
  Grade 4: Life-threatening consequences; urgent intervention indicated. Grade 5: Death related to AE.
Time Frame: Day 1 to end of follow-up, up to a maximum of 60 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Part: 0.3 mg/kg | Dose Escalation Part: 0.6 mg/kg | Dose Escalation Part: 0.9 mg/kg | Dose Escalation Part: 1.2 mg/kg | Dose Escalation Part: 1.5 mg/kg | Dose Escalation Part: 1.8 mg/kg | Dose Escalation Part: 2.0 mg/kg | Dose Escalation Part: 2.2 mg/kg | Dose Expansion Part: Bladder Cancer | Dose Expansion Part: Cervical Cancer | Dose Expansion Part: Endometrial Cancer | Dose Expansion Part: Esophageal Cancer | Dose Expansion Part: Non-Small Cell Lung Cancer (NSCLC) | Dose Expansion Part: Ovarian Cancer | Dose Expansion Part: Prostate Cancer
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 15 | 55 | 14 | 15 | 15 | 36 | 18
Participants | 2 | 1 | 1 | 0 | 2 | 2 | 0 | 1 | 0 | 23 | 0 | 3 | 1 | 5 | 3

3. Secondary Outcome: Dose Escalation and Expansion Parts: Number of Participants With Markedly Abnormal Coagulation Values
Description: Number of participants with markedly abnormal coagulation values was defined as all participants who experienced at least 1 CTCAE grade >= 3 coagulation value.
  A markedly abnormal coagulation value was determined using the CTCAE grading systems based on National Cancer Institute (NCI)-CTCAE version 4.03 assessed by the investigator per the below definitions.
  Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living.
  Grade 4: Life-threatening consequences; urgent intervention indicated. Grade 5: Death related to AE.
Time Frame: Day 1 to end of follow-up, up to a maximum of 60 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Part: 0.3 mg/kg | Dose Escalation Part: 0.6 mg/kg | Dose Escalation Part: 0.9 mg/kg | Dose Escalation Part: 1.2 mg/kg | Dose Escalation Part: 1.5 mg/kg | Dose Escalation Part: 1.8 mg/kg | Dose Escalation Part: 2.0 mg/kg | Dose Escalation Part: 2.2 mg/kg | Dose Expansion Part: Bladder Cancer | Dose Expansion Part: Cervical Cancer | Dose Expansion Part: Endometrial Cancer | Dose Expansion Part: Esophageal Cancer | Dose Expansion Part: Non-Small Cell Lung Cancer (NSCLC) | Dose Expansion Part: Ovarian Cancer | Dose Expansion Part: Prostate Cancer
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 15 | 55 | 14 | 15 | 15 | 36 | 18
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 7 | 2 | 0 | 2 | 5 | 4

4. Secondary Outcome: Dose Escalation and Expansion Part: Number of Participants With Markedly Abnormal Biochemistry Values
Description: Number of participants with markedly abnormal biochemistry results were defined as all participants who experienced at least 1 CTCAE grade >= 3 biochemistry value.
  A markedly abnormal biochemistry value was determined using the CTCAE grading systems based on National Cancer Institute (NCI)-CTCAE version 4.03 assessed by the investigator per the below definitions.
  Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living.
  Grade 4: Life-threatening consequences; urgent intervention indicated. Grade 5: Death related to AE.
Time Frame: Day 1 to end of follow-up, up to a maximum of 60 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Part: 0.3 mg/kg | Dose Escalation Part: 0.6 mg/kg | Dose Escalation Part: 0.9 mg/kg | Dose Escalation Part: 1.2 mg/kg | Dose Escalation Part: 1.5 mg/kg | Dose Escalation Part: 1.8 mg/kg | Dose Escalation Part: 2.0 mg/kg | Dose Escalation Part: 2.2 mg/kg | Dose Expansion Part: Bladder Cancer | Dose Expansion Part: Cervical Cancer | Dose Expansion Part: Endometrial Cancer | Dose Expansion Part: Esophageal Cancer | Dose Expansion Part: Non-Small Cell Lung Cancer (NSCLC) | Dose Expansion Part: Ovarian Cancer | Dose Expansion Part: Prostate Cancer
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 15 | 55 | 14 | 15 | 15 | 36 | 18
Participants | 2 | 1 | 3 | 0 | 1 | 0 | 1 | 2 | 4 | 8 | 4 | 6 | 2 | 9 | 4

5. Secondary Outcome: Dose Escalation and Expansion Parts: Number of Participants Who Experienced a Skin Rash
Time Frame: Day 1 to end of follow-up, up to a maximum of 60 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Part: 0.3 mg/kg | Dose Escalation Part: 0.6 mg/kg | Dose Escalation Part: 0.9 mg/kg | Dose Escalation Part: 1.2 mg/kg | Dose Escalation Part: 1.5 mg/kg | Dose Escalation Part: 1.8 mg/kg | Dose Escalation Part: 2.0 mg/kg | Dose Escalation Part: 2.2 mg/kg | Dose Expansion Part: Bladder Cancer | Dose Expansion Part: Cervical Cancer | Dose Expansion Part: Endometrial Cancer | Dose Expansion Part: Esophageal Cancer | Dose Expansion Part: Non-Small Cell Lung Cancer (NSCLC) | Dose Expansion Part: Ovarian Cancer | Dose Expansion Part: Prostate Cancer
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 15 | 55 | 14 | 15 | 15 | 36 | 18
Participants | 1 | 0 | 0 | 2 | 0 | 2 | 2 | 4 | 3 | 6 | 2 | 2 | 2 | 8 | 5

6. Secondary Outcome: Dose Escalation and Expansion Parts: Number of Participants Who Experienced a Bleeding Event of Special Interest
Description: Bleeding adverse events of special interest included treatment emergent adverse events with preferred terms within the following standardised MedDRA queries (SMQs): Haemorrhage terms, excluding laboratory terms SMQ [20000039] (Broad) and Haemorrhage, laboratory terms SMQ [20000040] (Narrow).
  Bleeding adverse events of special interest were evaluated according to the NCI-CTCAE version 4.03. Bleeding events of all grades are included.
  Grade 1:Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living.
  Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living.
  Grade 4: Life-threatening consequences; urgent intervention indicated. Grade 5: Death related to AE.
Time Frame: Day 1 to end of follow-up, up to a maximum of 60 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Part: 0.3 mg/kg | Dose Escalation Part: 0.6 mg/kg | Dose Escalation Part: 0.9 mg/kg | Dose Escalation Part: 1.2 mg/kg | Dose Escalation Part: 1.5 mg/kg | Dose Escalation Part: 1.8 mg/kg | Dose Escalation Part: 2.0 mg/kg | Dose Escalation Part: 2.2 mg/kg | Dose Expansion Part: Bladder Cancer | Dose Expansion Part: Cervical Cancer | Dose Expansion Part: Endometrial Cancer | Dose Expansion Part: Esophageal Cancer | Dose Expansion Part: Non-Small Cell Lung Cancer (NSCLC) | Dose Expansion Part: Ovarian Cancer | Dose Expansion Part: Prostate Cancer
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 15 | 55 | 14 | 15 | 15 | 36 | 18
Participants | 0 | 1 | 0 | 3 | 3 | 3 | 2 | 5 | 10 | 31 | 10 | 7 | 9 | 27 | 10

7. Secondary Outcome: Dose Escalation and Expansion Part: Number of Participants Who Experienced a Peripheral Neuropathy Event
Description: Peripheral neuropathy events of special interest were evaluated according to the NCI-CTCAE version 4.03. Peripheral neuropathy events of all grades are included in the numbers below.
  Grade 1:Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living.
  Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living.
  Grade 4: Life-threatening consequences; urgent intervention indicated. Grade 5: Death related to AE.
Time Frame: Day 1 to end of follow-up, up to a maximum of 60 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Part: 0.3 mg/kg | Dose Escalation Part: 0.6 mg/kg | Dose Escalation Part: 0.9 mg/kg | Dose Escalation Part: 1.2 mg/kg | Dose Escalation Part: 1.5 mg/kg | Dose Escalation Part: 1.8 mg/kg | Dose Escalation Part: 2.0 mg/kg | Dose Escalation Part: 2.2 mg/kg | Dose Expansion Part: Bladder Cancer | Dose Expansion Part: Cervical Cancer | Dose Expansion Part: Endometrial Cancer | Dose Expansion Part: Esophageal Cancer | Dose Expansion Part: Non-Small Cell Lung Cancer (NSCLC) | Dose Expansion Part: Ovarian Cancer | Dose Expansion Part: Prostate Cancer
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 15 | 55 | 14 | 15 | 15 | 36 | 18
Participants | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 5 | 17 | 6 | 3 | 5 | 17 | 7

8. Secondary Outcome: Dose Escalation Part: Clearance of Tisotumab Vedotin and Total HuMax-TF
Description: Pharmacokinetic (PK) parameters in plasma were determined based on non compartmental methods and calculated separately for Cycle 1 and Cycle 2 in each part of the study. Data was not collected to report or calculate clearance for the expansion phase.
Time Frame: Before infusion, Day 1 (pre-dose) and 0.25 to 336 hours post-dose of Cycle 1 and Cycle 2 (each cycle was 21 days)
Population: PK analysis set: all participants who had been exposed to tisotumab vedotin and had at least 1 PK assessment after first dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hr/kg
Arm/Group | Dose Escalation Part: 0.3 mg/kg | Dose Escalation Part: 0.6 mg/kg | Dose Escalation Part: 0.9 mg/kg | Dose Escalation Part: 1.2 mg/kg | Dose Escalation Part: 1.5 mg/kg | Dose Escalation Part: 1.8 mg/kg | Dose Escalation Part: 2.0 mg/kg | Dose Escalation Part: 2.2 mg/kg
Number analyzed (Participants) | 0 | 3 | 3 | 3 | 3 | 3 | 3 | 5
mL/hr/kg
  Tisotumab Vedotin: Cycle 1 |  | 1.61 (7.79) | 1.46 (15.23) | 1.07 (11.60) | 1.84 (20.59) | 1.17 (60.05) | 1.56 (34.12) | 0.87 (8.93)
  Tisotumab Vedotin: Cycle 2: number analyzed (Participants) | 0 | 2 | 3 | 3 | 3 | 2 | 2 | 3
  Tisotumab Vedotin: Cycle 2 |  | 1.72 (4.98) | 1.44 (6.32) | 1.07 (10.45) | 2.05 (26.80) | 0.93 (24.03) | 1.30 (19.06) | 1.03 (11.34)
  Total HuMax-TF: Cycle 1: number analyzed (Participants) | 0 | 2 | 3 | 3 | 3 | 3 | 3 | 5
  Total HuMax-TF: Cycle 1 |  | 1.02 (0.20) | 0.98 (16.90) | 0.69 (12.61) | 1.26 (31.29) | 0.81 (69.72) | 0.87 (33.85) | 0.56 (14.13)
  Total HuMax-TF: Cycle 2: number analyzed (Participants) | 0 | 2 | 3 | 3 | 3 | 2 | 2 | 3
  Total HuMax-TF: Cycle 2 |  | 1.05 (9.95) | 0.98 (6.52) | 0.71 (13.41) | 1.40 (31.39) | 0.53 (12.41) | 0.82 (26.45) | 0.61 (9.72)

9. Secondary Outcome: Dose Escalation Part: Volume of Distribution of Tisotumab Vedotin and Total HuMax-TF
Description: PK parameters in plasma were determined based on non compartmental methods and calculated separately for Cycle 1 and Cycle 2 in each part of the study. Data was not planned to be collected for the volume of distribution of tisotumab vedotin and total HuMax-TF for the dose expansion part.
Time Frame: Before infusion, Day 1 (pre-dose) and 0.25 to 336 hours post-dose of Cycle 1 and Cycle 2 (each cycle was 21 days)
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/kg
Arm/Group | Dose Escalation Part: 0.3 mg/kg | Dose Escalation Part: 0.6 mg/kg | Dose Escalation Part: 0.9 mg/kg | Dose Escalation Part: 1.2 mg/kg | Dose Escalation Part: 1.5 mg/kg | Dose Escalation Part: 1.8 mg/kg | Dose Escalation Part: 2.0 mg/kg | Dose Escalation Part: 2.2 mg/kg
Number analyzed (Participants) | 0 | 3 | 3 | 3 | 3 | 3 | 3 | 5
mL/kg
  Tisotumab Vedotin: Cycle 1 |  | 68.40 (11.84) | 70.80 (14.54) | 63.46 (16.87) | 86.10 (12.38) | 81.13 (35.60) | 92.04 (21.62) | 61.46 (18.07)
  Tisotumab Vedotin: Cycle 2: number analyzed (Participants) | 0 | 2 | 3 | 3 | 3 | 2 | 2 | 3
  Tisotumab Vedotin: Cycle 2 |  | 76.69 (9.53) | 69.74 (7.99) | 62.61 (6.03) | 99.20 (20.82) | 70.21 (42.93) | 74.82 (4.19) | 72.74 (5.79)
  Total HuMax-TF: Cycle 1: number analyzed (Participants) | 0 | 2 | 3 | 3 | 3 | 3 | 3 | 5
  Total HuMax-TF: Cycle 1 |  | 51.55 (1.61) | 60.27 (17.79) | 57.38 (8.65) | 77.55 (10.74) | 67.26 (50.61) | 68.69 (30.52) | 50.69 (7.20)
  Total HuMax-TF: Cycle 2: number analyzed (Participants) | 0 | 2 | 3 | 3 | 3 | 2 | 2 | 3
  Total HuMax-TF: Cycle 2 |  | 55.75 (10.80) | 57.13 (8.90) | 58.48 (12.66) | 84.98 (22.85) | 50.62 (36.02) | 60.40 (17.48) | 58.10 (12.31)

10. Secondary Outcome: Dose Escalation and Expansion Part: Area Under the Curve From Time Zero to the Last Measurable Concentration (AUC0-t) of Tisotumab Vedotin and Total HuMax-TF
Description: PK parameters in plasma were determined based on non-compartmental methods and calculated separately for Cycle 1 and Cycle 2 in each part of the study.
Time Frame: Before infusion, Day 1 (pre-dose) and 0.25 to 336 hours post-dose of Cycle 1 and Cycle 2 (each cycle was 21 days)
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/mL
Groups:
- Dose Expansion Part: Pharmacokinetics (PK) Analysis Set: PK was only planned to be analyzed per the dose level received, not per cancer type. So the PK data is pooled for all participants in the dose expansion part of the study.
Arm/Group | Dose Escalation Part: 0.3 mg/kg | Dose Escalation Part: 0.6 mg/kg | Dose Escalation Part: 0.9 mg/kg | Dose Escalation Part: 1.2 mg/kg | Dose Escalation Part: 1.5 mg/kg | Dose Escalation Part: 1.8 mg/kg | Dose Escalation Part: 2.0 mg/kg | Dose Escalation Part: 2.2 mg/kg | Dose Expansion Part: Pharmacokinetics (PK) Analysis Set
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 168
day*ug/mL
  Tisotumab Vedotin: Cycle 1: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 167
  Tisotumab Vedotin: Cycle 1 | 2.5 (3.1) | 15.4 (8.2) | 25.1 (16.9) | 45.2 (9.3) | 33.1 (19.0) | 63.0 (49.3) | 52.3 (33.1) | 84.9 (33.7) | 79.31 (49.40)
  Tisotumab Vedotin: Cycle 2: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 146
  Tisotumab Vedotin: Cycle 2 | 2.0 (15.7) | 9.9 (49.1) | 25.6 (7.1) | 45.2 (10.1) | 29.8 (25.1) | 42.7 (72.7) | 62.7 (21.5) | 86.3 (14.4) | 68.54 (55.49)
  Total HuMax-TF: Cycle 1 | 2.9 (0.5) | 15.4 (53.1) | 35.0 (18.9) | 60.4 (13.4) | 44.9 (27.8) | 86.7 (54.3) | 85.9 (36.7) | 123.0 (34.7) | 112.70 (45.23)
  Total HuMax-TF: Cycle 2: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 146
  Total HuMax-TF: Cycle 2 | 2.4 (12.3) | 14.4 (55.4) | 35.7 (7.1) | 58.8 (15.5) | 40.9 (26.2) | 60.2 (76.6) | 92.5 (33.4) | 133.6 (13.9) | 114.54 (45.83)

11. Secondary Outcome: Dose Escalation Part: Area Under the Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Tisotumab Vedotin and Total HuMax-TF
Description: PK parameters in plasma were determined based on non compartmental methods and calculated separately for Cycle 1 and Cycle 2. AUC0-inf was only analyzed in the dose escalation part of the study. Data was not planned to be collected for the AUC0-inf of tisotumab vedotin and total HuMax-TF for the dose expansion part.
Time Frame: Before infusion, Day 1 (pre-dose) and 0.25 to 336 hours post-dose of Cycle 1 and Cycle 2 (each cycle was 21 days)
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/mL
Arm/Group | Dose Escalation Part: 0.3 mg/kg | Dose Escalation Part: 0.6 mg/kg | Dose Escalation Part: 0.9 mg/kg | Dose Escalation Part: 1.2 mg/kg | Dose Escalation Part: 1.5 mg/kg | Dose Escalation Part: 1.8 mg/kg | Dose Escalation Part: 2.0 mg/kg | Dose Escalation Part: 2.2 mg/kg
Number analyzed (Participants) | 0 | 3 | 3 | 3 | 3 | 3 | 3 | 6
day*ug/mL
  Tisotumab Vedotin: Cycle 1 |  | 15.57 (7.81) | 25.77 (15.70) | 46.68 (10.99) | 33.95 (20.93) | 63.88 (48.61) | 53.47 (30.88) | 105.84 (8.68)
  Tisotumab Vedotin: Cycle 2: number analyzed (Participants) | 0 | 3 | 3 | 3 | 3 | 2 | 2 | 3
  Tisotumab Vedotin: Cycle 2 |  | 14.52 (4.98) | 26.12 (6.44) | 46.59 (9.98) | 30.56 (26.43) | 80.59 (24.03) | 64.10 (19.06) | 88.95 (11.04)
  Total HuMax-TF: Cycle 1: number analyzed (Participants) | 0 | 2 | 3 | 3 | 3 | 3 | 3 | 2
  Total HuMax-TF: Cycle 1 |  | 23.75 (0.20) | 37.02 (16.39) | 69.96 (13.26) | 48.19 (35.67) | 90.08 (52.74) | 93.29 (30.45) | 157.81 (12.70)
  Total HuMax-TF: Cycle 2: number analyzed (Participants) | 0 | 2 | 3 | 3 | 3 | 2 | 2 | 3
  Total HuMax-TF: Cycle 2 |  | 23.01 (9.95) | 37.08 (6.37) | 67.93 (14.25) | 43.41 (30.31) | 136.08 (12.41) | 98.59 (26.45) | 145.82 (9.42)

12. Secondary Outcome: Dose Escalation and Expansion Part: Maximum Observed Plasma Concentration (Cmax) of Tisotumab Vedotin and Total HuMax-TF
Description: as for outcome 10
Time Frame: Before infusion, Day 1 (pre-dose) and 0.25 to 336 hours post-dose of Cycle 1 and Cycle 2 (each cycle was 21 days)
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Dose Escalation Part: 0.3 mg/kg | Dose Escalation Part: 0.6 mg/kg | Dose Escalation Part: 0.9 mg/kg | Dose Escalation Part: 1.2 mg/kg | Dose Escalation Part: 1.5 mg/kg | Dose Escalation Part: 1.8 mg/kg | Dose Escalation Part: 2.0 mg/kg | Dose Escalation Part: 2.2 mg/kg | Dose Expansion Part: Pharmacokinetics (PK) Analysis Set
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 168
ug/mL
  Tisotumab Vedotin: Cycle 1: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 167
  Tisotumab Vedotin: Cycle 1 | 4.78 (12.35) | 12.20 (9.47) | 19.81 (17.32) | 34.67 (18.48) | 23.12 (21.10) | 35.42 (39.20) | 32.30 (22.08) | 55.53 (10.31) | 29.1 (34.1)
  Tisotumab Vedotin: Cycle 2: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 146
  Tisotumab Vedotin: Cycle 2 | 3.85 (27.65) | 12.51 (11.51) | 20.25 (5.14) | 32.38 (7.11) | 21.84 (24.97) | 35.92 (30.39) | 44.30 (0.32) | 48.79 (26.37) | 26.1 (41.2)
  Total HuMax-TF: Cycle 1 | 4.90 (13.00) | 11.84 (8.31) | 17.98 (11.64) | 29.30 (10.14) | 23.55 (25.16) | 30.57 (37.42) | 38.78 (21.77) | 58.02 (12.77) | 39.8 (31.1)
  Total HuMax-TF: Cycle 2: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 146
  Total HuMax-TF: Cycle 2 | 3.96 (21.83) | 11.54 (8.83) | 16.90 (1.57) | 31.33 (8.13) | 22.11 (21.03) | 37.71 (42.96) | 43.40 (6.67) | 53.67 (19.75) | 38.3 (33.3)

13. Secondary Outcome: Dose Escalation and Expansion Part: Time of Cmax (Tmax) of Tisotumab Vedotin and Total HuMax-TF
Description: as for outcome 10
Time Frame: Before infusion, Day 1 (pre-dose) and 0.25 to 336 hours post-dose of Cycle 1 and Cycle 2 (each cycle was 21 days)
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Dose Escalation Part: 0.3 mg/kg | Dose Escalation Part: 0.6 mg/kg | Dose Escalation Part: 0.9 mg/kg | Dose Escalation Part: 1.2 mg/kg | Dose Escalation Part: 1.5 mg/kg | Dose Escalation Part: 1.8 mg/kg | Dose Escalation Part: 2.0 mg/kg | Dose Escalation Part: 2.2 mg/kg | Dose Expansion Part: Pharmacokinetics (PK) Analysis Set
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 168
hours
  Tisotumab Vedotin: Cycle 1: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 167
  Tisotumab Vedotin: Cycle 1 | 1.47 (72.74) | 1.18 (13.03) | 1.34 (11.77) | 1.15 (11.66) | 1.12 (9.55) | 1.18 (14.30) | 1.18 (7.45) | 1.11 (12.52) | 1.21 (364.12)
  Tisotumab Vedotin: Cycle 2: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 146
  Tisotumab Vedotin: Cycle 2 | 1.54 (63.29) | 1.34 (6.27) | 1.32 (5.96) | 1.13 (11.18) | 1.21 (16.61) | 2.44 (35.75) | 1.14 (9.29) | 1.29 (7.55) | 1.44 (303.89)
  Total HuMax-TF: Cycle 1 | 2.20 (49.15) | 1.18 (13.03) | 1.34 (11.77) | 1.15 (11.66) | 1.12 (9.55) | 1.18 (14.30) | 1.18 (7.45) | 1.11 (12.52) | 1.10 (397.92)
  Total HuMax-TF: Cycle 2: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 146
  Total HuMax-TF: Cycle 2 | 2.19 (46.56) | 1.34 (6.27) | 1.32 (5.96) | 1.13 (11.18) | 1.21 (16.61) | 1.76 (50.43) | 1.14 (9.29) | 1.29 (7.55) | 1.15 (356.23)

14. Secondary Outcome: Dose Escalation Part: Half-life (t1/2) of Tisotumab Vedotin and Total HuMax-TF
Description: PK parameters in plasma were determined based on non-compartmental methods and calculated separately for Cycle 1 and Cycle 2. t1/2 was only analyzed for the dose escalation part of the study. Data was not planned to be collected for t1/2 of tisotumab vedotin and total HuMax-TF for the dose expansion part.
Time Frame: Before infusion, Day 1 (pre-dose) and 0.25 to 336 hours post-dose of Cycle 1 and Cycle 2 (each cycle was 21 days)
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Dose Escalation Part: 0.3 mg/kg | Dose Escalation Part: 0.6 mg/kg | Dose Escalation Part: 0.9 mg/kg | Dose Escalation Part: 1.2 mg/kg | Dose Escalation Part: 1.5 mg/kg | Dose Escalation Part: 1.8 mg/kg | Dose Escalation Part: 2.0 mg/kg | Dose Escalation Part: 2.2 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6
hours
  Tisotumab Vedotin: Cycle 1 | 12.22 (11.61) | 29.53 (4.08) | 33.72 (6.26) | 41.06 (6.85) | 32.42 (20.05) | 47.89 (25.82) | 40.93 (11.48) | 41.19 (34.02)
  Tisotumab Vedotin: Cycle 2: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 2 | 2 | 3
  Tisotumab Vedotin: Cycle 2 | 13.54 (5.50) | 23.50 (39.89) | 33.68 (1.74) | 40.44 (4.69) | 33.62 (14.50) | 32.15 (62.74) | 39.89 (23.15) | 48.93 (5.61)
  Total HuMax-TF: Cycle 1: number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 6
  Total HuMax-TF: Cycle 1 | 16.05 (27.93) | 28.66 (30.64) | 42.52 (7.48) | 57.37 (8.65) | 42.72 (34.62) | 57.72 (17.47) | 54.95 (5.32) | 55.10 (27.36)
  Total HuMax-TF: Cycle 2: number analyzed (Participants) | 3 | 2 | 3 | 3 | 3 | 2 | 2 | 3
  Total HuMax-TF: Cycle 2 | 18.34 (8.73) | 30.71 (27.65) | 40.37 (4.27) | 56.77 (9.60) | 42.18 (25.39) | 46.24 (53.11) | 51.06 (9.18) | 66.05 (10.07)

15. Secondary Outcome: Dose Escalation and Expansion Part: AUC0-t of Free Monomethyl Auristatin E (MMAE)
Description: PK parameters in plasma were determined based on non compartmental methods and calculated separately for Cycle 1 and Cycle 2 in each part of the study.
Time Frame: Before infusion, Day 1 (pre-dose) and 0.25 to 336 hours post-dose of Cycle 1 and Cycle 2 (each cycle was 21 days)
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ng/mL
Arm/Group | Dose Escalation Part: 0.3 mg/kg | Dose Escalation Part: 0.6 mg/kg | Dose Escalation Part: 0.9 mg/kg | Dose Escalation Part: 1.2 mg/kg | Dose Escalation Part: 1.5 mg/kg | Dose Escalation Part: 1.8 mg/kg | Dose Escalation Part: 2.0 mg/kg | Dose Escalation Part: 2.2 mg/kg | Dose Expansion Part: Pharmacokinetics (PK) Analysis Set
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 168
day*ng/mL
  Cycle 1 | 6.20 (72.05) | 12.61 (28.18) | 12.22 (67.23) | 11.63 (52.69) | 26.55 (44.24) | 22.55 (57.26) | 67.42 (59.98) | 26.47 (59.35) | 25.80 (93.91)
  Cycle 2: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 145
  Cycle 2 | 3.19 (140.85) | 4.69 (87.27) | 14.89 (66.97) | 16.92 (58.12) | 21.51 (34.25) | 18.97 (52.14) | 36.20 (33.82) | 37.50 (43.08) | 23.48 (76.47)

16. Secondary Outcome: Dose Escalation Part: AUC0-inf of Free MMAE
Description: PK parameters in plasma were determined based on non-compartmental methods and calculated separately for Cycle 1 and Cycle 2. AUC0-inf was not planned to be collected for the dose expansion part. AUC0-inf was not calculated where the percentage of the AUC that was due to the extrapolation was more than 20%.
Time Frame: Before infusion, Day 1 (pre-dose) and 0.25 to 336 hours post-dose of Cycle 1 and Cycle 2 (each cycle was 21 days)
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ng/mL
Arm/Group | Dose Escalation Part: 0.3 mg/kg | Dose Escalation Part: 0.6 mg/kg | Dose Escalation Part: 0.9 mg/kg | Dose Escalation Part: 1.2 mg/kg | Dose Escalation Part: 1.5 mg/kg | Dose Escalation Part: 1.8 mg/kg | Dose Escalation Part: 2.0 mg/kg | Dose Escalation Part: 2.2 mg/kg
Number analyzed (Participants) | 2 | 1 | 2 | 1 | 2 | 1 | 1 | 1
day*ng/mL
  Cycle 1 | 12.63 (12.44) | 13.93 (NA) — Only 1 participant had evaluable data, so geometric coefficient of variation could not be calculated. | 16.32 (57.56) | 20.39 (NA) — Only 1 participant had evaluable data, so geometric coefficient of variation could not be calculated. | 27.08 (58.96) | 25.29 (NA) — Only 1 participant had evaluable data, so geometric coefficient of variation could not be calculated. | 78.31 (NA) — Only 1 participant had evaluable data, so geometric coefficient of variation could not be calculated. | 63.03 (NA) — Only 1 participant had evaluable data, so geometric coefficient of variation could not be calculated.
  Cycle 2: number analyzed (Participants) | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 1
  Cycle 2 |  |  | 22.32 (43.62) | 31.40 (NA) — Only 1 participant had evaluable data, so geometric coefficient of variation could not be calculated. | 31.43 (NA) — Only 1 participant had evaluable data, so geometric coefficient of variation could not be calculated. | 33.23 (NA) — Only 1 participant had evaluable data, so geometric coefficient of variation could not be calculated. |  | 58.95 (NA) — Only 1 participant had evaluable data, so geometric coefficient of variation could not be calculated.

17. Secondary Outcome: Dose Escalation and Expansion Part: Cmax of Free MMAE
Description: as for outcome 10
Time Frame: Before infusion, Day 1 (pre-dose) and 0.25 to 336 hours post-dose of Cycle 1 and Cycle 2 (each cycle was 21 days)
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dose Escalation Part: 0.3 mg/kg | Dose Escalation Part: 0.6 mg/kg | Dose Escalation Part: 0.9 mg/kg | Dose Escalation Part: 1.2 mg/kg | Dose Escalation Part: 1.5 mg/kg | Dose Escalation Part: 1.8 mg/kg | Dose Escalation Part: 2.0 mg/kg | Dose Escalation Part: 2.2 mg/kg | Dose Expansion Part: Pharmacokinetics (PK) Analysis Set
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 168
ng/mL
  Cycle 1 | 0.760 (62.505) | 1.673 (30.756) | 1.524 (54.491) | 1.410 (19.149) | 2.807 (39.398) | 2.587 (29.172) | 6.351 (61.505) | 4.877 (31.350) | 3.16 (88.30)
  Cycle 2: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 145
  Cycle 2 | 1.091 (74.293) | 1.342 (24.320) | 2.059 (51.470) | 2.243 (50.367) | 2.718 (39.492) | 2.035 (39.785) | 3.369 (36.875) | 4.704 (18.856) | 2.73 (78.69)

18. Secondary Outcome: Dose Escalation and Expansion Part: Tmax of Free MMAE
Description: as for outcome 10
Time Frame: Before infusion, Day 1 (pre-dose) and 0.25 to 336 hours post-dose of Cycle 1 and Cycle 2 (each cycle was 21 days)
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Dose Escalation Part: 0.3 mg/kg | Dose Escalation Part: 0.6 mg/kg | Dose Escalation Part: 0.9 mg/kg | Dose Escalation Part: 1.2 mg/kg | Dose Escalation Part: 1.5 mg/kg | Dose Escalation Part: 1.8 mg/kg | Dose Escalation Part: 2.0 mg/kg | Dose Escalation Part: 2.2 mg/kg | Dose Expansion Part: Pharmacokinetics (PK) Analysis Set
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 168
hours
  Cycle 1 | 23.88 (4.41) | 22.77 (16.56) | 24.39 (7.72) | 24.19 (5.52) | 25.07 (0.68) | 47.74 (114.28) | 83.24 (67.57) | 84.88 (61.54) | 154.28 (54.214)
  Cycle 2: number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 145
  Cycle 2 | 23.73 (5.78) | 24.05 (8.48) | 23.92 (13.04) | 24.94 (1.48) | 25.26 (0.76) | 46.24 (112.48) | 65.15 (104.61) | 47.12 (112.10) | 125.38 (31.21)

19. Secondary Outcome: Dose Escalation Part: PK Parameters, T 1/2 of Free MMAE
Description: PK parameters in plasma were determined based on non compartmental methods and calculated separately for Cycle 1 and Cycle 2. T1/2 was determined only for the dose escalation part of the study.
Time Frame: Before infusion, Day 1 (pre-dose) and 0.25 to 336 hours post-dose of Cycle 1 and Cycle 2 (each cycle was 21 days)
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Dose Escalation Part: 0.3 mg/kg | Dose Escalation Part: 0.6 mg/kg | Dose Escalation Part: 0.9 mg/kg | Dose Escalation Part: 1.2 mg/kg | Dose Escalation Part: 1.5 mg/kg | Dose Escalation Part: 1.8 mg/kg | Dose Escalation Part: 2.0 mg/kg | Dose Escalation Part: 2.2 mg/kg
Number analyzed (Participants) | 2 | 1 | 2 | 1 | 2 | 1 | 1 | 1
hours
  Cycle 1 | 95.15 (25.74) | 69.34 (NA) — Only 1 participant had evaluable data, so geometric coefficient of variation could not be calculated. | 63.98 (2.24) | 62.58 (NA) — Only 1 participant had evaluable data, so geometric coefficient of variation could not be calculated. | 63.65 (7.86) | 78.90 (NA) — Only 1 participant had evaluable data, so geometric coefficient of variation could not be calculated. | 57.74 (NA) — Only 1 participant had evaluable data, so geometric coefficient of variation could not be calculated. | 68.47 (NA) — Only 1 participant had evaluable data, so geometric coefficient of variation could not be calculated.
  Cycle 2: number analyzed (Participants) | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 1
  Cycle 2 |  |  | 69.65 (3.86) | 60.71 (NA) — Only 1 participant had evaluable data, so geometric coefficient of variation could not be calculated. | 70.20 (NA) — Only 1 participant had evaluable data, so geometric coefficient of variation could not be calculated. | 78.94 (NA) — Only 1 participant had evaluable data, so geometric coefficient of variation could not be calculated. |  | 63.92 (NA) — Only 1 participant had evaluable data, so geometric coefficient of variation could not be calculated.

20. Secondary Outcome: Dose Escalation and Expansion Part: Number of Participants With Positive Anti-Drug Antibodies (ADAs) to Tisotumab Vedotin
Description: Participants who met the criterion for positive ADAs on treatment were defined as participants who were negative at baseline and had at least one positive post-baseline result, or participants who were positive at baseline and had at least one post baseline result with a titer higher than baseline.
Time Frame: Day 1 to end of follow-up, up to a maximum of 60 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Part: 0.3 mg/kg | Dose Escalation Part: 0.6 mg/kg | Dose Escalation Part: 0.9 mg/kg | Dose Escalation Part: 1.2 mg/kg | Dose Escalation Part: 1.5 mg/kg | Dose Escalation Part: 1.8 mg/kg | Dose Escalation Part: 2.0 mg/kg | Dose Escalation Part: 2.2 mg/kg | Dose Expansion Part: Bladder Cancer | Dose Expansion Part: Cervical Cancer | Dose Expansion Part: Endometrial Cancer | Dose Expansion Part: Esophageal Cancer | Dose Expansion Part: Non-Small Cell Lung Cancer (NSCLC) | Dose Expansion Part: Ovarian Cancer | Dose Expansion Part: Prostate Cancer
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 15 | 55 | 14 | 15 | 15 | 36 | 18
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 1

21. Secondary Outcome: Dose Escalation Part: Anti-Tumor Activity Measured by Number of Participants Who Experienced Tumor Shrinkage
Description: Anti-tumor activity measured by the number of participants who experienced tumor shrinkage was not planned to be collected for the dose expansion part.
Time Frame: Day 1 to end of follow-up, up to a maximum of 60 weeks
Population: Full analysis set: all participants who had been exposed to tisotumab vedotin in the dose escalation part.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Part: 0.3 mg/kg | Dose Escalation Part: 0.6 mg/kg | Dose Escalation Part: 0.9 mg/kg | Dose Escalation Part: 1.2 mg/kg | Dose Escalation Part: 1.5 mg/kg | Dose Escalation Part: 1.8 mg/kg | Dose Escalation Part: 2.0 mg/kg | Dose Escalation Part: 2.2 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6
Participants | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 3

22. Primary Outcome: Dose Expansion Part: Evaluation of Treatment-Emergent Adverse Events
Description: Evaluation of treatment-emergent adverse events (TEAEs) includes number of participants with at least one:
  TEAE Serious TEAE Infusion-related TEAE Common Terminology Criteria for Adverse Events (CTCAE) grade >=3 Treatment-related TEAE
  A CTCAE TEAE was determined using the CTCAE grading systems based on NCI-CTCAE version 4.03 assessed by the investigator per the below definitions.
  Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living.
  Grade 4: Life-threatening consequences; urgent intervention indicated. Grade 5: Death related to AE.
Time Frame: Treatment emergent adverse events are reported from Day 1 to 30 days after dosing. The treatment duration ranged from 1 to 325 days in the dose expansion part.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Expansion Part: Bladder Cancer | Dose Expansion Part: Cervical Cancer | Dose Expansion Part: Endometrial Cancer | Dose Expansion Part: Esophageal Cancer | Dose Expansion Part: Non-Small Cell Lung Cancer (NSCLC) | Dose Expansion Part: Ovarian Cancer | Dose Expansion Part: Prostate Cancer
Number analyzed (Participants) | 15 | 55 | 14 | 15 | 15 | 36 | 18
Participants
  TEAEs | 15 | 55 | 14 | 15 | 15 | 36 | 18
  Serious TEAEs | 7 | 26 | 5 | 8 | 6 | 13 | 6
  Infusion-Related TEAEs | 1 | 1 | 1 | 1 | 2 | 0 | 0
  CTCAE Grade >=3 TEAEs | 9 | 30 | 8 | 8 | 10 | 16 | 11
  TEAEs Related to Study Drug | 15 | 54 | 13 | 14 | 14 | 36 | 18

23. Secondary Outcome: Dose Expansion Part: Anti-Tumor Activity Measured by Maximum Reduction Among Available Post-Baseline Sum of Lesion Measurements
Description: Anti-tumor activity measured by maximum reduction among available post-baseline sum of lesion measurements was not planned to be collected for the dose escalation part.
Time Frame: Day 1 to end of follow-up, up to a maximum of 60 weeks
Population: The number of participants analyzed includes all participants with baseline and one post-baseline evaluable tumor assessment
Measure: Median (Full Range); unit: millimeter(s)
Arm/Group | Dose Expansion Part: Bladder Cancer | Dose Expansion Part: Cervical Cancer | Dose Expansion Part: Endometrial Cancer | Dose Expansion Part: Esophageal Cancer | Dose Expansion Part: Non-Small Cell Lung Cancer (NSCLC) | Dose Expansion Part: Ovarian Cancer | Dose Expansion Part: Prostate Cancer
Number analyzed (Participants) | 14 | 50 | 12 | 11 | 14 | 33 | 12
millimeter(s) | 6.00 [-127.0 to 41.0] | -8.50 [-64.0 to 50.0] | 1.00 [-11.0 to 26.0] | -2.00 [-51.0 to 40.0] | 0.00 [-59.0 to 31.0] | -4.00 [-41.0 to 115.0] | -1.00 [-11.0 to 15.0]

24. Secondary Outcome: Dose Escalation and Expansion Part: Percentage Change From Baseline in Prostate Specific Antigen (PSA)
Description: PSA was only assessed in participants with castrate-resistant prostate cancer.
Time Frame: Day 1 to end of follow-up, up to a maximum of 60 weeks
Population: Analyses includes all participants with castrate-resistant prostate cancer who have a baseline and end of study evaluable assessment.
Measure: Median (Full Range); unit: Percentage Change in PSA
Arm/Group | Dose Escalation Part: 0.3 mg/kg | Dose Escalation Part: 0.6 mg/kg | Dose Escalation Part: 0.9 mg/kg | Dose Escalation Part: 1.2 mg/kg | Dose Escalation Part: 1.5 mg/kg | Dose Escalation Part: 1.8 mg/kg | Dose Escalation Part: 2.0 mg/kg | Dose Escalation Part: 2.2 mg/kg | Dose Expansion Part: Prostate Cancer
Number analyzed (Participants) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 11
Percentage Change in PSA |  | 64.35 [64.35 to 64.35] |  | 40.91 [40.91 to 40.91] | 3.92 [3.92 to 3.92] |  |  |  | 60.07 [3.4 to 996.5]

25. Secondary Outcome: Dose Escalation and Expansion Part: Percentage Change From Baseline in CA-125
Description: In the dose escalation part, CA-125 was only assessed for participants with ovarian cancer. In the dose expansion part, CA-125 was intended to be assessed only for participants with ovarian and endometrium cancer, but was additionally assessed for some participants with NSCLC and cervical cancer.
Time Frame: Day 1 to end of follow-up, up to a maximum of 60 weeks
Population: Analyses includes all participants in the dose escalation and expansion parts with ovarian cancer and some participants with NSCLC and cervical cancer in the dose expansion part who have a baseline and end of study evaluable assessment.
Measure: Median (Full Range); unit: Percentage Change
Groups:
- Dose Expansion Part: Cervical Cancer: Participants with cervical cancer received tisotumab vedotin on Day 1 of each cycle (each treatment cycle was 21 days) as an IV infusion at a dose of 2.0mg/kg of body weight.
Arm/Group | Dose Escalation Part: 0.3 mg/kg | Dose Escalation Part: 0.6 mg/kg | Dose Escalation Part: 0.9 mg/kg | Dose Escalation Part: 1.2 mg/kg | Dose Escalation Part: 1.5 mg/kg | Dose Escalation Part: 1.8 mg/kg | Dose Escalation Part: 2.0 mg/kg | Dose Escalation Part: 2.2 mg/kg | Dose Expansion Part: Cervical Cancer | Dose Expansion Part: Endometrial Cancer | Dose Expansion Part: Non-Small Cell Lung Cancer (NSCLC) | Dose Expansion Part: Ovarian Cancer
Number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 8 | 10 | 3 | 25
Percentage Change |  |  |  | 18.75 [18.75 to 18.75] |  | -13.98 [-13.98 to -13.98] | 113.71 [113.71 to 113.71] | 11.62 [-22.7 to 45.9] | -25.17 [-88.7 to 240.5] | 37.85 [-46.1 to 666.2] | 180.94 [47.1 to 980.5] | 73.19 [-89.0 to 1924.4]

26. Secondary Outcome: Dose Escalation and Expansion Part: Objective Response Rate
Description: Objective Response Rate per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. Response assessment was investigator based for the escalation part and Independent Review Committee (IRC) based for the expansion part.
Time Frame: Day 1 to end of follow-up, up to a maximum of 60 weeks
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Dose Escalation Part: 0.3 mg/kg | Dose Escalation Part: 0.6 mg/kg | Dose Escalation Part: 0.9 mg/kg | Dose Escalation Part: 1.2 mg/kg | Dose Escalation Part: 1.5 mg/kg | Dose Escalation Part: 1.8 mg/kg | Dose Escalation Part: 2.0 mg/kg | Dose Escalation Part: 2.2 mg/kg | Dose Expansion Part: Bladder Cancer | Dose Expansion Part: Cervical Cancer | Dose Expansion Part: Endometrial Cancer | Dose Expansion Part: Esophageal Cancer | Dose Expansion Part: Non-Small Cell Lung Cancer (NSCLC) | Dose Expansion Part: Ovarian Cancer | Dose Expansion Part: Prostate Cancer
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 15 | 55 | 14 | 15 | 15 | 36 | 18
Percentage of Participants | 0 [0 to 71] | 0 [0 to 71] | 0 [0 to 71] | 33 [1 to 91] | 0 [0 to 71] | 0 [0 to 71] | 0 [0 to 71] | 0 [0 to 46] | 27 [8 to 55] | 24 [13 to 37] | 7 [0 to 34] | 13 [2 to 40] | 13 [2 to 40] | 14 [5 to 29] | 0 [0 to 19]

27. Secondary Outcome: Dose Escalation and Expansion Part: Disease Control Rate
Description: Disease control rate was defined as the percentage of participants with CR, PR or stable disease (SD) as per investigator assessment per RECIST version 1.1 after 6, 12, 24 and 36 weeks. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for Progressive Disease.
Time Frame: At 6, 12, 24 and 36 weeks
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Dose Escalation Part: 0.3 mg/kg | Dose Escalation Part: 0.6 mg/kg | Dose Escalation Part: 0.9 mg/kg | Dose Escalation Part: 1.2 mg/kg | Dose Escalation Part: 1.5 mg/kg | Dose Escalation Part: 1.8 mg/kg | Dose Escalation Part: 2.0 mg/kg | Dose Escalation Part: 2.2 mg/kg | Dose Expansion Part: Bladder Cancer | Dose Expansion Part: Cervical Cancer | Dose Expansion Part: Endometrial Cancer | Dose Expansion Part: Esophageal Cancer | Dose Expansion Part: Non-Small Cell Lung Cancer (NSCLC) | Dose Expansion Part: Ovarian Cancer | Dose Expansion Part: Prostate Cancer
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 15 | 55 | 14 | 15 | 15 | 36 | 18
Percentage of Participants
  Week 6 | 0 [0 to 71] | 33 [1 to 91] | 33 [1 to 91] | 67 [9 to 99] | 33 [1 to 91] | 100 [29 to 100] | 67 [9 to 99] | 50 [12 to 88] | 47 [21 to 73] | 60 [46 to 73] | 64 [35 to 87] | 40 [16 to 68] | 60 [32 to 84] | 72 [55 to 86] | 61 [36 to 83]
  Week 12 | 0 [0 to 71] | 33 [1 to 91] | 33 [1 to 91] | 67 [9 to 99] | 0 [0 to 71] | 67 [9 to 99] | 33 [1 to 91] | 0 [0 to 46] | 33 [12 to 62] | 47 [34 to 61] | 43 [18 to 71] | 20 [4 to 48] | 13 [2 to 40] | 42 [26 to 59] | 28 [10 to 53]
  Week 24 | 0 [0 to 71] | 33 [1 to 91] | 0 [0 to 71] | 33 [1 to 91] | 0 [0 to 71] | 0 [0 to 71] | 0 [0 to 71] | 0 [0 to 46] | 20 [4 to 48] | 18 [9 to 31] | 21 [5 to 51] | 7 [0 to 32] | 13 [2 to 40] | 14 [5 to 29] | 6 [0 to 27]
  Week 36 | 0 [0 to 71] | 33 [1 to 91] | 0 [0 to 71] | 33 [1 to 91] | 0 [0 to 71] | 0 [0 to 71] | 0 [0 to 71] | 0 [0 to 46] | 7 [0 to 32] | 11 [4 to 22] | 0 [0 to 23] | 0 [0 to 22] | 7 [0 to 32] | 3 [0 to 15] | 6 [0 to 27]

28. Secondary Outcome: Dose Escalation and Expansion Part: Progression Free Survival (PFS)
Description: PFS was defined as the time in weeks from Day 1 in Cycle 1 to first disease progression or death, whichever occurred earliest, as assessed by the investigator. Only deaths that occurred within 60 days of the last visit were considered in the analysis and result are presented based on Kaplan-Meier estimates. Progression as defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase from nadir in the sum of diameters of target lesions, unequivocal progression in non-target lesions, or the appearance of new lesions
Time Frame: Day 1 to end of follow-up, up to a maximum of 60 weeks
Population: Participants with documented disease progression and/or death are included.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Dose Escalation Part: 0.3 mg/kg | Dose Escalation Part: 0.6 mg/kg | Dose Escalation Part: 0.9 mg/kg | Dose Escalation Part: 1.2 mg/kg | Dose Escalation Part: 1.5 mg/kg | Dose Escalation Part: 1.8 mg/kg | Dose Escalation Part: 2.0 mg/kg | Dose Escalation Part: 2.2 mg/kg | Dose Expansion Part: Bladder Cancer | Dose Expansion Part: Cervical Cancer | Dose Expansion Part: Endometrial Cancer | Dose Expansion Part: Esophageal Cancer | Dose Expansion Part: Non-Small Cell Lung Cancer (NSCLC) | Dose Expansion Part: Ovarian Cancer | Dose Expansion Part: Prostate Cancer
Number analyzed (Participants) | 3 | 3 | 2 | 2 | 3 | 2 | 3 | 3 | 10 | 41 | 4 | 10 | 9 | 26 | 12
Weeks | 5.1 [4.9 to 5.4] | 6.0 [3.9 to 49.1] | 6.1 [4.9 to NA] — Upper limit was not estimable because of insufficient number of participants with events prior to censoring. | 27.1 [6.0 to NA] — Upper limit was not estimable because of insufficient number of participants with events prior to censoring. | 6.1 [5.3 to 10.4] | 17.1 [11.3 to NA] — Upper limit was not estimable because of insufficient number of participants with events prior to censoring | 12.3 [5.0 to 14.1] | 11.3 [2.1 to 11.3] | 11.0 [5.1 to 43.0] | 18.1 [9.3 to 23.0] | NA [5.1 to NA] — Median and upper limit were not estimable because of insufficient number of participants with events prior to censoring. | 10.1 [5.3 to 17.0] | 13.0 [5.1 to 17.3] | 13.0 [12.1 to 18.3] | 12.9 [7.1 to 23.7]

29. Secondary Outcome: Dose Expansion Part: Duration of Response (DOR)
Description: DOR was defined as the median time in weeks from when confirmed response was first documented until the first documented disease progression, or death from any cause, whichever was earliest as assessed by the investigator. A responder was defined as any participant with a best overall response of confirmed CR or PR.
Time Frame: Day 1 to end of follow-up, up to a maximum of 60 weeks
Population: All participants who had a confirmed response of either CR or PR and were considered a responder for the study.
Measure: Median (95% Confidence Interval); unit: Weeks
Groups:
- Dose Escalation Part: 0.3 mg/kg: Dose Escalation Part: 0.3 mg/kgEdit Participants received tisotumab vedotin on Day 1 of each cycle (each treatment cycle was 21 days) as an intravenous (IV) infusion at a dose of 0.3 mg/kg of body weight.
- Dose Escalation Part: 0.6 mg/kg: Dose Escalation Part: 0.6 mg/kgEdit Participants received tisotumab vedotin on Day 1 of each cycle (each treatment cycle was 21 days) as an IV infusion at a dose of 0.6 mg/kg of body weight.
- Dose Escalation Part: 0.9 mg/kg: Dose Escalation Part: 0.9 mg/kgEdit Participants received tisotumab vedotin on Day 1 of each cycle (each treatment cycle was 21 days) as an IV infusion at a dose of 0.9 mg/kg of body weight.
Arm/Group | Dose Escalation Part: 0.3 mg/kg | Dose Escalation Part: 0.6 mg/kg | Dose Escalation Part: 0.9 mg/kg | Dose Escalation Part: 1.2 mg/kg | Dose Escalation Part: 1.5 mg/kg | Dose Escalation Part: 1.8 mg/kg | Dose Escalation Part: 2.0 mg/kg | Dose Escalation Part: 2.2 mg/kg | Dose Expansion Part: Bladder Cancer | Dose Expansion Part: Cervical Cancer | Dose Expansion Part: Endometrial Cancer | Dose Expansion Part: Esophageal Cancer | Dose Expansion Part: Non-Small Cell Lung Cancer (NSCLC) | Dose Expansion Part: Ovarian Cancer | Dose Expansion Part: Prostate Cancer
Number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 13 | 1 | 2 | 2 | 5 | 0
Weeks |  |  |  | NA [NA to NA] — Duration of response could not be estimated because DOR was censored for the single responder. |  |  |  |  | 32.0 [11.0 to 32.0] | 18.4 [13.1 to 41.7] | NA [NA to NA] — Duration of response could not be estimated because DOR was censored for the single responder. | 18.3 [11.6 to 25.0] | NA [12.0 to NA] — Duration of response and the upper CI limit could not be estimated because DOR for one responder was censored later than the observed DOR for the other responder. | 21.4 [13.1 to 29.6] |

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events are reported from Day 1 to 30 days after dosing. The treatment duration ranged from 1 to 249 days in the escalation part and from 1 to 325 days in the expansion part.
Description: Deaths from all causes are reported from day of enrollment to end of follow up (up to maximum of 60 weeks).
Groups:
- Dose Expansion Part: Non-Small-Cell Lung Cancer: Participants with NSCLC received tisotumab vedotin on Day 1 of each cycle (each treatment cycle was 21 days) as an IV infusion at a dose of 2.0 mg/kg of body weight.
Arm/Group | Dose Escalation Part: 0.3 mg/kg | Dose Escalation Part: 0.6 mg/kg | Dose Escalation Part: 0.9 mg/kg | Dose Escalation Part: 1.2 mg/kg | Dose Escalation Part: 1.5 mg/kg | Dose Escalation Part: 1.8 mg/kg | Dose Escalation Part: 2.0 mg/kg | Dose Escalation Part: 2.2 mg/kg | Dose Expansion Part: Bladder Cancer | Dose Expansion Part: Cervical Cancer | Dose Expansion Part: Endometrial Cancer | Dose Expansion Part: Esophageal Cancer | Dose Expansion Part: Non-Small-Cell Lung Cancer | Dose Expansion Part: Ovarian Cancer | Dose Expansion Part: Prostate Cancer
All-Cause Mortality (participants affected / at risk) | 2/3 | 1/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/6 | 0/15 | 2/55 | 0/14 | 1/15 | 1/15 | 2/36 | 1/18
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 0/3 | 2/3 | 2/3 | 2/3 | 2/3 | 4/6 | 7/15 | 26/55 | 5/14 | 8/15 | 6/15 | 13/36 | 6/18
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 6/6 | 15/15 | 55/55 | 14/14 | 15/15 | 15/15 | 36/36 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation Part: 0.3 mg/kg (N=3) | Dose Escalation Part: 0.6 mg/kg (N=3) | Dose Escalation Part: 0.9 mg/kg (N=3) | Dose Escalation Part: 1.2 mg/kg (N=3) | Dose Escalation Part: 1.5 mg/kg (N=3) | Dose Escalation Part: 1.8 mg/kg (N=3) | Dose Escalation Part: 2.0 mg/kg (N=3) | Dose Escalation Part: 2.2 mg/kg (N=6) | Dose Expansion Part: Bladder Cancer (N=15) | Dose Expansion Part: Cervical Cancer (N=55) | Dose Expansion Part: Endometrial Cancer (N=14) | Dose Expansion Part: Esophageal Cancer (N=15) | Dose Expansion Part: Non-Small-Cell Lung Cancer (N=15) | Dose Expansion Part: Ovarian Cancer (N=36) | Dose Expansion Part: Prostate Cancer (N=18)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Micrococcus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis escherichia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Klebsiella infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Guillain-barre syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stent malfunction (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular disorders (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation Part: 0.3 mg/kg (N=3) | Dose Escalation Part: 0.6 mg/kg (N=3) | Dose Escalation Part: 0.9 mg/kg (N=3) | Dose Escalation Part: 1.2 mg/kg (N=3) | Dose Escalation Part: 1.5 mg/kg (N=3) | Dose Escalation Part: 1.8 mg/kg (N=3) | Dose Escalation Part: 2.0 mg/kg (N=3) | Dose Escalation Part: 2.2 mg/kg (N=6) | Dose Expansion Part: Bladder Cancer (N=15) | Dose Expansion Part: Cervical Cancer (N=55) | Dose Expansion Part: Endometrial Cancer (N=14) | Dose Expansion Part: Esophageal Cancer (N=15) | Dose Expansion Part: Non-Small-Cell Lung Cancer (N=15) | Dose Expansion Part: Ovarian Cancer (N=36) | Dose Expansion Part: Prostate Cancer (N=18)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Contrast media allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Conjunctival scar (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelid contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharynx radiation injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chemical burns of eye (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intermittent claudication (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urine flow decreased (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 5 (7) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (3) | 1 (3) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 7 (7) | 25 (30) | 7 (8) | 7 (8) | 10 (16) | 20 (30) | 12 (14)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (2) | 3 (3) | 6 (7) | 19 (21) | 3 (3) | 6 (8) | 5 (5) | 11 (13) | 9 (11)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 3 (3) | 17 (26) | 6 (8) | 2 (4) | 4 (4) | 14 (19) | 5 (7)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 18 (23) | 4 (6) | 4 (5) | 6 (6) | 11 (18) | 6 (9)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 15 (17) | 1 (1) | 1 (1) | 2 (2) | 8 (9) | 6 (8)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 4 (4) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 5 (6) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 6 (7) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal mucosal hyperplasia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (3) | 3 (4) | 2 (2) | 4 (5) | 13 (13) | 28 (40) | 11 (13) | 8 (10) | 11 (15) | 30 (34) | 12 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 8 (8) | 3 (3) | 2 (2) | 3 (3) | 6 (7) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 5 (8) | 1 (1) | 3 (3) | 5 (5) | 3 (3) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 1 (1) | 4 (6) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 6 (6) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 3 (3) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal crusting (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 4 (4) | 8 (10) | 29 (34) | 10 (12) | 10 (10) | 8 (11) | 15 (18) | 15 (16)
Pyrexia (General disorders) | 2 (4) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 11 (13) | 1 (1) | 2 (3) | 0 (0) | 4 (5) | 0 (0)
Mucosal inflammation (General disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 5 (5) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 5 (5) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (7) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (5) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Influenza like illness (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 4 (4) | 3 (3) | 22 (22) | 8 (8) | 4 (4) | 7 (7) | 19 (19) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (5) | 10 (11) | 2 (3) | 2 (3) | 1 (1) | 6 (7) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 7 (8) | 4 (4) | 1 (1) | 2 (2) | 6 (6) | 4 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 4 (4) | 4 (5) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 5 (6) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 7 (9) | 23 (37) | 6 (8) | 4 (5) | 6 (7) | 15 (19) | 9 (9)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 2 (3) | 2 (3) | 11 (16) | 0 (0) | 1 (1) | 0 (0) | 4 (6) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemophilus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urethritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 16 (19) | 5 (5) | 2 (2) | 3 (3) | 10 (12) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 5 (5) | 2 (3) | 0 (0) | 1 (1) | 9 (9) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (7) | 3 (3) | 1 (1) | 1 (2) | 5 (6) | 3 (3)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Central pain syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amputation stump pain (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 3 (3) | 20 (22) | 5 (6) | 6 (7) | 5 (5) | 12 (13) | 10 (14)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 11 (14) | 1 (2) | 2 (2) | 2 (2) | 5 (6) | 2 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (6) | 1 (1) | 2 (3) | 0 (0) | 4 (4) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 5 (6) | 0 (0) | 2 (2) | 1 (1) | 9 (9) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 6 (6) | 2 (2) | 0 (0) | 2 (2) | 6 (7) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (3) | 6 (7) | 2 (2) | 1 (1) | 2 (2) | 3 (3) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 0 (0) | 1 (1) | 3 (4) | 4 (5) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 1 (2) | 2 (2) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis climacteric (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 14 (14) | 6 (6) | 2 (2) | 6 (7) | 6 (6) | 2 (2)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (3) | 5 (5) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 6 (6) | 0 (0)
Conjunctival ulcer (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Meibomianitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Noninfective conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Symblepharon (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ulcerative keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Foreign body sensation in eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Punctate keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Chorioretinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Open angle glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal vein occlusion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye inflammation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 4 (4) | 9 (10) | 4 (4) | 2 (2) | 2 (2) | 3 (3) | 6 (6)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 6 (9) | 3 (5) | 3 (3) | 2 (2) | 2 (2) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 7 (8) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 2 (2) | 0 (0) | 1 (2)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vital dye staining cornea present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival staining (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood fibrinogen increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serum ferritin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urea decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibrin d dimer increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 13 (17) | 2 (2) | 3 (4) | 2 (2) | 0 (0) | 3 (6)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 6 (6) | 2 (2) | 1 (1) | 4 (4) | 6 (7) | 2 (2)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All proposed publications and presentations shall be submitted to the sponsor for its review at least 30 days before such presentation or publication is submitted to any third party.

DOCUMENTS (2):
  • Study Protocol (2018-07-18): https://cdn.clinicaltrials.gov/large-docs/23/NCT02001623/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/23/NCT02001623/SAP_001.pdf